CLINICAL TRIAL: NCT02838212
Title: Adverse Drug Reactions With Fatal Outcome
Status: Completed | Type: Observational
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Eva Montané, Clinical Pharmacologist, Germans Trias i Pujol Hospital
Other Study IDs: RAM-MORT 2015
Record Dates: First submitted 2016-07-13; First posted 2016-07-20 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Adverse Drug Reaction
Keywords: adverse drug reaction; hospital mortality; incidence
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions | interventions — Adverse Drug Reaction Reporting Systems; Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Drug-related deaths: fatal adverse drug reactions
  Interventions: Drug: adverse drug reaction
- non drug-related deaths: deaths for other causes different as drugs

INTERVENTIONS:
Drug: adverse drug reaction — drug-related death
  Other Names: side effect
  Groups: Drug-related deaths

SUMMARY:
The purpose of this study is to determine the incidence of drug-related deaths in a university hospital during the year 2015

DETAILED DESCRIPTION:
The investigators aimed to determine the incidence of drug-related mortality of admitted patients in a university hospital during the year 2015

ELIGIBILITY:
Inclusion Criteria:

* inpatients deaths and drug-related deaths.

Exclusion Criteria:

* death patients in the emergency room, patients with a death diagnosis not available, and dead patients due to other causes non-drug related.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All inpatients dead in the Germans Trias i Pujol University Hospital during the year 2015.
  Patients with a death diagnosis in a predefined list of medical conditions, potentially caused by drugs, were the selected cases for further review.
Sampling Method: Non-Probability Sample
Enrollment: 1135 (Actual)
Dates: Start 2016-02; Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Incidence of drug-related deaths of all hospital admissions | during the year 2015

SECONDARY OUTCOMES:
Number of drug-related deaths with the suspected drug started the previous week | during the year 2015
Number of drug-related deaths with drug interactions between suspected drugs | during the year 2015
Number of preventable drug-related deaths assessed by Schumock criteria | during the year 2015
Number of drug-related deaths with polypharmacy | during the year 2015
  Polypharmacy: when patient received >10 drugs
Number of drug-related deaths with autopsy | during the year 2015
Number of drug-related deaths in which the suspected drug had a contributive role | during the year 2015
Number of drug-related deaths with "certain" or "probable" categories assessed by World Health Organization (WHO) criteria and Naranjo algorithm | during the year 2015
Number of drug-related deaths presented during hospitalization | during the year 2015
Risk factors of drug-related deaths | during the year 2015
  risk factors assessed: age, sex, Charlson score, and hospitalization length
Incidence of drug-related deaths of all inpatients deaths | during the year 2015.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Montané, PhD, Principal Investigator — Department of Clinical Pharmacology. Hospital Universitari Germans Trias i Pujol. Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No